CLINICAL TRIAL: NCT05427903
Title: Evaluation of Two Approaches in Enhancing the Efficacy of Inferior Alveolar Nerve Block During Treatment of Mandibular First Permanent Molars With Symptomatic Irreversible Pulpitis: A Randomized Parallel Controlled Trial
Brief Title: Two Approaches in Enhancing the Efficacy of Inferior Alveolar Nerve Block During Treatment of Mandibular First Permanent Molars With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 602
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural | interventions — Cryotherapy; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryotherapy (Experimental)
  Interventions: Procedure: Buccal local anesthetic infiltration using articaine 4% 1:100000 epinephrine
- IANB plus buccal infiltration local anesthesia (Experimental)
  Interventions: Procedure: Cryotherapy
- IANB (Active Comparator)
  Interventions: Procedure: Cryotherapy; Procedure: Buccal local anesthetic infiltration using articaine 4% 1:100000 epinephrine

INTERVENTIONS:
Procedure: Cryotherapy — Ice packs application for 5 minutes after IANB injection
  Arms: IANB; IANB plus buccal infiltration local anesthesia
Procedure: Buccal local anesthetic infiltration using articaine 4% 1:100000 epinephrine — Buccal infiltration after IANB
  Arms: Cryotherapy; IANB

SUMMARY:
The study is designed as a randomized parallel controlled trial with three groups. Participants aged above 18 years with the first permanent molars with symptomatic signs of irreversible pulpitis will be randomly assigned into 3 groups. The first group (experimental group) will be injected with 4% articaine 1:100.000 epinephrine (inferior alveolar nerve block) will be anesthetized using 4% articaine 1:100.000 plus cryotherapy application, and the second group (experimental group) will be anaesthetised with IANB plus buccal infiltration. For the third group (control group), the mandibular molars will be anaesthetized using epinephrine using the inferior alveolar nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years
* Presence of at least one mandibular first permanent molar, with signs and symptoms of irreversible pulpititis

Exclusion Criteria:

* Participants with a history of taking medications that could interfere with the action of the anaesthetic solutions
* Presence of paresthesia
* Presence of psychological problems
* Taking analgesics or other medications that would alter the inflammatory response of the pulp or provide analgesia 12 h pre-operatively

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-06-18 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | up to 24 hours
  verbal rating scale (VRS) withh the following scores: Score 0: no pain, Score 1: mild pain, Score 2: moderate pain, and Score 3: severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt